#### **CONSENT TO TAKE PART IN RESEARCH**

#### Dartmouth College

Children's multimedia study Diane Gilbert-Diamond, ScD

<u>Introduction</u>: You and your child are being asked to take part in a research study. Taking part in research is voluntary.

You and your child are being asked to take part in this study because your child meets the age requirement for the study and is interested in participating in the study.

Your and your child's decision whether or not to take part will not influence your and your child's future medical care, job status, academic standing, etc. Please ask questions if there is anything about this study you do not understand.

#### What is the purpose of this study?

The purpose of the study is to investigate the impact of media multi-tasking, the process of simultaneously attending to multiple electronic media devices, on food-related behaviors in children. Common examples of media multi-tasking include 1) texting while watching TV and 2) surfing the internet while talking on the phone. One of the main questions that we are addressing is how media multi-tasking impacts the amount of attention children give to food cues, as well as the effect the media multi-tasking has on snacking behavior.

### Will you and your child benefit from taking part in this study?

You and your child will not personally benefit from being in this research study. We hope to gather information that may help people in the future.

## What does this study involve?

Your and your child's participation in this study involves three 1-hour visits to the lab, with each visit one to three weeks apart. During the visit(s):

- Your child may eat some foods.
- Your child may answer simple questions.
- Your child may play some computer games while having their eyes tracked using an eye tracker. There will not be any object placed on your child's eyes. The eye tracker is a screen-based device that uses a high-resolution camera mounted to the bottom of a monitor to track where a person is looking on the screen. It is non-invasive and does not require any equipment to be placed on the head, or around the eye. It records where a person is looking by recording

a video of the participant's eye movements. Critically, the video used to track the eyes is not saved.

- You may complete some online questionnaires.
- We may measure your child's height and weight.

In between the first and second visit, your child may be asked to wear an activity monitor (like a fitbit) for several days, and you will be asked to help him/her keep the monitor on and keep a log.

## What are the options if you/your child do/does not want to take part in this study?

The alternative is not to take part in this study.

#### If you take part in this study, what activities will be done only for research purposes?

All the procedures, tests, and activities described in this consent form are being done only for research purposes.

#### What are the risks involved with taking part in this study?

Although the risk involved in this study is minimal, children with food allergies could experience adverse reactions to food served. In order to prevent allergic reactions, *please inform us of any food allergies your child has*. Children with severe food allergies may not take part in this study.

| Food(s) your child is alle | rgic to (write N/A if your child has none): |
|----------------------------|---------------------------------------------|
| Severity and symptoms: | |

## Other important items you should know:

- Leaving the study: You may choose to stop taking part in this study at any time for any reason. If you decide to stop taking part, it will have no effect on your and your child's future medical care, job status, academic standing, etc.
- **New Information:** New information related to this research will be made known to you when it becomes available. This may affect your decision to stay in this study.
- **Funding:** Dartmouth College is the sponsor of this research. They provided funding for this research.
- **Number of people in this study:** We expect up to 150 children to enroll in this study.

## How will your privacy be protected?

For this study, we may collect your and your child's health behavior and sociodemographic information. We are careful to protect the identities of people in this study. We will keep all study information secure and confidential. All collected data will be de-identified with random number

v. 11/20/2019

coding, and only the principal investigators and the research team members who directly contact the participants will have access to the information necessary to link them to their de-identified data. The encrypted database on a secure Dartmouth server will be password-protected. All paper files will be stored in a locked file cabinet in a secure office. When the data are no longer needed, electronic data will be permanently deleted from the database, and paper files will be securely shredded and destroyed.

The information collected for this study will be used only for purposes of the research as stated earlier in this form. Please note that the HIPAA Privacy Rule does not recognize as valid any authorization for the use or disclosure of Protected Health Information (PHI) for future, unspecified research projects.

#### Who may use or see your child's health information?

By signing this form, you allow the research team to use your child's health information and give it to others involved in the research. The research team includes the study director plus others working on this study at Dartmouth-Hitchcock Medical Center and elsewhere. You also permit any health care provider holding your child's height and weight information needed for this study to give this information to the research team.

The information collected for this study may be used by researchers or officials of the following institutions.

- Dartmouth College
- Mary Hitchcock Memorial Hospital
- Dartmouth-Hitchcock Clinic
- Dartmouth-Hitchcock Medical Center
- Other collaborating research institutions

In order to conduct this study, researchers need to use your child's health care information. Although no information is being gathered from your child's medical record, and no information is being added to the medical record as part of this study- the information created as part of this study is considered Protected Health Information ("PHI"). PHI is protected by federal privacy laws (HIPAA). By signing this consent form, you give your permission to have your child's PHI collected, used and disclosed for purposes of this study. There is no intention to disclose your child's PHI to others outside of the study. There are protections in place to keep your child's PHI and research data confidential. However, HIPAA requires notification so you are aware *if your child's* PHI is disclosed to others, it may no longer be protected by federal privacy laws.

No publication or public presentation about the research described above will reveal your child's identity without another authorization from you.

Identifiable data collected for this study will be used for research purposes which are determined to

v. 11/20/2019

be reasonable and in line with expectations by a review committee.

Once data collected for this research study is no longer identifiable, the data may be used or disclosed for other purposes.

Your permission to use your child's health information for this study will not end until the study is completed. During this study, your child and others who take part in the study may not have access to the study data. You may ask for study data once the study is over. You have a right to receive a copy of the information in your child's medical record at any time.

It is possible for a court or government official to order the release of study data including information about your child.

# What if you decide not to give permission to use and share your child's personal health information?

If you do not allow use of your child's health information for this study, your child may not take part in this study.

If you or your child choose to stop taking part in this study, you may cancel permission for the use of your child's health information. You should let the researcher know if you want to cancel your permission. The study team will assist you in putting your wishes in writing. Information collected for the study before your permission is cancelled will continue to be used in the research.

# Will you be paid to take part in this study?

Your child will receive \$30 for the first visit, \$40 for the second visit, and \$70 for the third visit for their participation. In addition, your child will receive \$20 for keeping the activity monitor on and keeping a log in between the first and second study visit. You will receive \$10 for completing the parent questionnaire. If you qualify for mileage reimbursement, you will receive \$10 for each visit. Please note that you may receive some or all compensation in the form of gift cards.

### Whom should you call with questions about this study?

If you have questions about this study, or to report a research problem, you can call your doctor or the research directors for this study: Dr. Diane Gilbert-Diamond at (603) 653-3362 during normal business hours.

If you have questions, concerns, complaints, or suggestions about human research at Dartmouth, you may call the Office of the Committee for the Protection of Human Subjects at Dartmouth College (603) 646-6482 during normal business hours.

## **CONSENT**

I have read the above information about Children's Multimedia Study and have been provided with contact information to ask any questions that I have. I agree to grant permission for my child to take part in this study and I will receive a confirmation email this electronically signed consent form for my records.

#### SIGNATURE OPTIONS

| Participant's Signature and Date | PRINTED NAME |
|-------------------------------------------|--------------|
| Researcher or Designee Signature and Date | PRINTED NAME |